CLINICAL TRIAL: NCT00422695
Title: Pain and Sensory Changes Assessment in HIV+ Patients, A Model for Pain and Sensory Changes Related Compromised Immune System.
Brief Title: Pain and Sensory Changes Assessment in HIV+ Patients
Status: Completed | Type: Observational
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120060172
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-01

CONDITIONS: HIV Infections
Keywords: HIV; Quantitative Sensory Testing; Neuropathy; Treatment Experienced; Treatment Naive
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV +: Groups divided according to CD4 counts
- Healthy Controls: HIV -ve subjects

SUMMARY:
There are about 42 million people in the world afflicted with HIV or AIDS with about 1 million patients in the US.

The epidemiology of orofacial pain has been reported extensively in the literature, yet the prevalence severity and level of pain affecting the head, face, neck and intraoral structures has not been explored in a population of HIV infected individuals.

Pain, in general terms, is a common experience in HIV infected patients, even in the absence of cancer or opportunistic infections. There is a variation in the prevalence of pain in these individuals depending on the stage of disease, care setting, and study methods. The purpose of this study is:

1. To investigate the prevalence of orofacial pain in HIV infected patients during routine dental clinical assessment.
2. To study the sensory phenotype of HIV+ patients and healthy volunteers using Quantitative Sensory Testing:

   * To detect the presence of sensory aberrations in the orofacial complex;
   * To identify which nerve types are involved;
   * To identify the type of orofacial pain based on both sensory testing and clinical findings.
3. To determine psychological condition and nutrition status in patients with HIV.
4. To find associations between inherited traits and development of neuropathic pain.

DETAILED DESCRIPTION:
Patients and control volunteers will be recruited from the Oral medicine Post-graduate clinic at NJDS. Medical history will be taken and will include age, gender, ethnicity, current and past illnesses, current and past medications, blood reports (CD4 and CD8 counts) which have been obtained during routine medical assessment. The clinician will perform a clinical head and neck examination. The examination shall include an extra-oral, cranial nerve and temporomandibular joint (TMJ) examination, and muscle palpation. A thorough intraoral examination will be performed. Patients will be examined for pathologies of the oral mucosa, teeth and periodontium prior to their participation in the study. The evaluation findings will be reported using the Research Diagnostic Criteria for Temperomandibular disorders. The patient will note level of pain on Visual Analogue Scale if there is any pre-existing orofacial pain. Psychological screening and nutritional questionnaires will be completed by the patient.

Quantitative Sensory Testing will be conducted bilaterally on the face and intraorally on the tongue. Extraorally, the infraorbital and mental nerves regions will be tested bilaterally using thermal and electrical detection thresholds. Intraorally the tongue will be tested bilaterally for thermal and electrical detection threshold.

Many of the differences among people in the way they respond to symptomatic therapies and their individual risk of HIV+ patients with neuropathic pain may be affected by their genetic makeup. We will search for these kinds of associations between inherited traits and development of neuropathic pain in this study.

If the patient presents with evidence for pathologies that requires extraction of any molar (based on clinical and radiographic findings), the patient will be assessed 3 days, 8 days post-extraction and then after 3 weeks for thermal and electrical detection thresholds.

Inclusion criteria:

Group I n = 40 HIV+ with CD4+T cells/mm³ > 500 as determined by previous routine medical examination and from previous blood reports.

Group II n = 40 HIV+ with CD4+T cells/mm³ 200-499 as determined by previous routine medical examination and from previous blood reports.

Group III n = 40 HIV+ with CD4+T cells/mm³ < 200 as determined by previous routine medical examination and from previous blood reports.

Control Group n = 40 Healthy with normal blood reports, without dental pathologies.

ELIGIBILITY:
Inclusion Criteria:

Group I n = 40 HIV+ with CD4+T cells/mm³ > 500 as determined by previous routine medical examination and from previous blood reports.

Group II n = 40 HIV+ with CD4+T cells/mm³ 200-499 as determined by previous routine medical examination and from previous blood reports.

Group III n = 40 HIV+ with CD4+T cells/mm³ < 200 as determined by previous routine medical examination and from previous blood reports.

Control Group n = 40 Healthy with normal blood reports, without dental pathologies.

Exclusion Criteria:

* Patients under 18 year of age.
* Pregnant women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV +ve subjects Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2007-01; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eli Eliav, DMD PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- New Jersey Dental School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV +: Groups divided according to CD4 counts 105 HIV subjects
- Healthy Controls: HIV -free subjects 38 Healthy Controls
Period: Overall Study
Arm/Group | HIV + | Healthy Controls
Started | 105 | 38
Completed | 105 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV + | Healthy Controls | Total
Number analyzed (Participants) | 105 | 38 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 38 | 143
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.97 (7.22) | 42.53 (12.57) | 45.06 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 14 | 56
  Male | 63 | 24 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 97 | 35 | 132
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 105 | 38 | 143

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Chronic Myogenic Pain, TMJ Disoder, and Burning Mouth Syndrome
Description: 1. To investigate the prevalence of orofacial pain in HIV infected patients during routine dental clinical assessment.
  To study the sensory phenotype of HIV+ patients and healthy volunteers using Quantitative Sensory Testing:
  * To detect the presence of sensory aberrations in the orofacial complex;
  * To identify which nerve types are involved;
  * To identify the type of orofacial pain based on both sensory testing and clinical findings.
    3.To determine psychological condition and nutrition status in patients with HIV.
    4.To find associations between inherited traits and development of neuropathic pain.
Time Frame: Tests were performed during regular clinical visit. The test duration was about an hour
Population: Comparisons of categorical variables were performed with Fischer's exact test. Trends in ordered categorical variables were tested with the chi square test.
Measure: Number; unit: Participants
Arm/Group | HIV + | Healthy Controls
Number analyzed (Participants) | 105 | 38
Participants
  Subjects with chronic Myogenic Pain | 72 | 8
  Subjects with TMJ Disorder | 37 | 7
  Subjects with Burning MouthSyndrome | 20 | 0

2. Primary Outcome: Spontaneous Pain Intensity
Description: Pain intensity as measured with Visual Analog Scale during the time of examination.
  The subjects were required to report their perceived level of pain on a 10 cm VAS scale from zero to 10 with zero being no pain and 10 representing the worst pain imaginable. Given the ease of use of this method and its current use to measure pain, VAS scales were adapted to measure patient perceived orofacial pain wherein subjects were asked to draw a vertical line at the point on the horizontal line which best represented their pain response. Where left 0 is no pain and right -10 is maximal pain.
Time Frame: The time of the examination
Population: Comparison was made between control and HIV+ subjects
Measure: Mean (Standard Deviation); unit: units on a scale (0 to 10)
Arm/Group | HIV + | Healthy Controls
Number analyzed (Participants) | 105 | 38
units on a scale (0 to 10)
  Pain in Orofacial Region | 2.13 (2.2) | 0.05 (0.3)
  Overall body pain | 3.69 (3.1) | 0.92 (1.9)
Statistical Analysis 1: Comparison: HIV + vs Healthy Controls; Test type: Superiority or Other; p < 0.05, Chi-squared
Statistical Analysis 2: Comparison: HIV + vs Healthy Controls; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse events were assessed during the examination. The patients were patients of records and were routinely examined in the clinic.
Description: No interventional procedures were made
Arm/Group | HIV + | Healthy Controls
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/38
Other Adverse Events (participants affected / at risk) | 0/105 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No